CLINICAL TRIAL: NCT00803361
Title: Duloxetine Versus Placebo in the Treatment of Patients With Generalized Anxiety Disorder in China
Brief Title: Duloxetine for the Treatment of Generalized Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11517; F1J-MC-HMFJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-12-03; First posted 2008-12-05 (Estimated); Results first posted 2010-12-17 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2010-11

CONDITIONS: Generalized Anxiety Disorder
Keywords: anxiety
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine (Experimental)
  Interventions: Drug: Duloxetine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — 60 to 120 mg, capsules, oral, once a day for 15 weeks
  Other Names: Cymbalta; LY248686
  Arms: Duloxetine
Drug: Placebo — placebo capsules, oral, once a day for 15 weeks
  Arms: Placebo

SUMMARY:
This is a 15 week study comparing how well duloxetine and placebo treatments improve generalized anxiety disorder

ELIGIBILITY:
Inclusion Criteria:

* Psychiatric Diagnosis of generalized anxiety disorder (GAD)
* Outpatients
* Meet Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnosis for GAD
* Clinical Global Impression (CGI) of Severity Score of at least moderate
* Sheehan Disability Scale (SDS) Global Functioning Impairment Score >= 12

Exclusion Criteria:

* Pregnancy or breast feeding
* Serious medical illness
* Other primary psychiatric diagnoses, such as major depressive disorder or substance abuse disorder within the past 6 months
* panic disorder, post-traumatic stress disorder (PTSD), or eating disorder in the last year
* lifetime history of bipolar or psychosis
* Any unstable serious medical condition for which duloxetine would not be allowed
* Any use of medications that are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2008-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time(UTC/GMT -5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- China (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kunming
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanjing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Xi'an

REFERENCES:
- [Derived] Wu WY, Wang G, Ball SG, Desaiah D, Ang QQ. Duloxetine versus placebo in the treatment of patients with generalized anxiety disorder in China. Chin Med J (Engl). 2011 Oct;124(20):3260-8. PMID 22088518

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Duloxetine | Placebo
Started | 108 | 102
Completed | 82 | 74
Not Completed | 26 | 28
Not completed — Adverse Event | 13 | 3
Not completed — Lack of Efficacy | 4 | 13
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 2 | 4
Not completed — Withdrawal by Subject | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Placebo | Total
Number analyzed (Participants) | 108 | 102 | 210
Age Continuous [Mean (Standard Deviation); unit: years] | 37.26 (11.85) | 38.02 (12.03) | 37.63 (11.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 56 | 106
  Male | 58 | 46 | 104
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 108 | 102 | 210
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 108 | 102 | 210

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Hospital Anxiety and Depression Scale (HADS) Anxiety Subscale Score at Endpoint
Description: A 14-item questionnaire with 2 subscales: anxiety and depression. Each item is rated on a 4-point scale, giving maximum scores of 21 for anxiety and depression. Scores of 11 or more on either subscale are considered to be a significant 'case' of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7, 'normal.'
Time Frame: Baseline, Week 15
Population: Participants with a baseline and at least one post-baseline result within each treatment group.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 107 | 100
Units on a scale
  Baseline | 12.76 (2.89) | 13.56 (2.96)
  Change from Baseline | -6.38 (4.44) | -5.29 (4.78)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.006, ANCOVA — p-value is for Change from Baseline; Change = Treatment + Pooled Investigator + Baseline; Mean Difference (Final Values) = -1.62, 95% CI 2-sided [-2.76 to -0.48]

2. Secondary Outcome: Change From Baseline in the Hamilton Anxiety (HAMA) Rating Scale Total Score at Endpoint
Description: The HAMA scale measures anxiety symptoms accompanying Major Depressive Disorder (MDD). Each item of the 14-item HAMA was scored from 0 (not present) to 4 (very severe), with a resulting maximum total score of 56.
Time Frame: Baseline, Week 15
Population: Participants with a baseline and at least one post-baseline result within each treatment group.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 107 | 100
Units on a scale
  Baseline | 24.50 (5.81) | 24.24 (5.16)
  Change from Baseline | -14.42 (9.05) | -11.62 (8.31)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.024, ANCOVA — p-value is for Change from Baseline; Change = Treatment + Pooled Investigator + Baseline; Mean Difference (Final Values) = -2.56, 95% CI 2-sided [-4.78 to -0.34]

3. Secondary Outcome: Mean Clinical Global Impressions (CGI) Improvement Score at Endpoint
Description: Measures clinician's perception of patient improvement at the time of assessment compared with the start of treatment. Scores range from 1 (very much better) to 7 (very much worse).
Time Frame: Week 15
Population: Participants with at least one post-baseline result within each treatment group.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 107 | 100
Units on a Scale | 2.08 (0.97) | 2.54 (1.20)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.004, ANOVA; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-0.74 to -0.15]

4. Secondary Outcome: Change From Baseline in Brief Pain Inventory (BPI) - Short Form Severity (BPI-S) and Interference (BPI-I) Scores at Endpoint
Description: BPI-S and BPI-I are self-reported scales measuring severity of pain and interference on function. Severity scores: 0 (no pain) to 10 (severe pain) on each question assessing worst pain, least pain, and average pain in past 24 hours, and pain right now. Interference scores: 0 (does not interfere) to 10 (completely interferes) on each question assessing interference of pain in past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life.
Time Frame: Baseline, Week 15
Population: Participants with a baseline and at least one post-baseline result within each treatment group.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 107 | 100
Units on a Scale
  Severity of Worst Pain Baseline | 3.39 (2.84) | 4.22 (3.03)
  Severity of Worst Pain Change | -1.78 (2.44) | -1.88 (2.78)
  Severity of Least Pain Baseline | 1.17 (1.51) | 1.51 (1.81)
  Severity of Least Pain Change | -0.67 (1.32) | -0.45 (1.70)
  Severity of Average Pain Baseline | 2.36 (2.26) | 2.77 (2.20)
  Severity of Average Pain Change | -1.25 (1.94) | -0.97 (2.06)
  Severity of Pain Right Now Baseline | 2.21 (2.58) | 2.30 (2.68)
  Severity of Pain Right Now Change | -1.41 (2.29) | -0.77 (2.54)
  Interference of Pain, General Activity, Baseline | 2.60 (2.81) | 2.66 (2.69)
  Interference of Pain, General Activity, Change | -1.43 (2.40) | -1.06 (2.43)
  Interference of Pain, Mood, Baseline | 2.97 (3.04) | 3.40 (2.87)
  Interference of Pain, Mood, Change | -1.49 (2.71) | -1.44 (2.57)
  Interference of Pain,Walking Ability, Baseline | 1.31 (2.07) | 1.56 (2.16)
  Interference of Pain,Walking Ability, Change | -0.63 (2.01) | -0.47 (1.95)
  Int. of Pain, Normal Work, Baseline | 2.53 (2.77) | 2.44 (2.67)
  Int. of Pain, Normal Work, Change | -1.25 (2.54) | -0.96 (2.43)
  Int. of Pain, Relations with Others, Baseline | 2.01 (2.59) | 2.01 (2.52)
  Int. of Pain, Relations with Others, Change | -1.07 (2.22) | -0.88 (2.07)
  Interference of Pain, Sleep, Baseline | 2.55 (3.09) | 3.23 (3.15)
  Interference of Pain, Sleep, Change | -1.16 (2.56) | -1.45 (2.68)
  Interference of Pain, Enjoyment of Life, Baseline | 2.51 (2.80) | 2.62 (2.37)
  Interference of Pain, Enjoyment of Life, Change | -1.27 (2.73) | -0.99 (2.20)
  Mean Interference Score, Baseline | 2.36 (2.46) | 2.56 (2.25)
  Mean Interference Score, Change | -1.18 (2.13) | -1.04 (1.84)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.125, ANCOVA — p-value is for Severity of Worst Pain Change; Change = Treatment + Pooled Investigator + Baseline; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.93 to 0.11]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.014, ANCOVA — p-value is for Severity of Least Pain Change; Change = Treatment + Pooled Investigator + Baseline; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.75 to -0.09]
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.012, ANCOVA — p-value is for Severity of Average Pain Change; Change = Treatment + Pooled Investigator + Baseline; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-0.93 to -0.11]
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA — p-value is for Severity of Pain Right Now Change; Change = Treatment + Pooled Investigator + Baseline; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-1.14 to -0.25]
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.101, ANCOVA — p-value is for Interference of Pain, General Activity, Change; Change = Treatment + Pooled Investigator + Baseline; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.87 to 0.08]
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.252, ANCOVA — p-value is for Interference of Pain, Mood, Change; Change = Treatment + Pooled Investigator + Baseline; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-0.83 to 0.22]
Statistical Analysis 7: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.149, ANCOVA — p-value is for Interference of Pain,Walking Ability, Change; Change = Treatment + Pooled Investigator + Baseline; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.72 to 0.11]
Statistical Analysis 8: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.367, ANCOVA — p-value is for Interference of Pain, Normal Work, Change; Change = Treatment + Pooled Investigator + Baseline; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.71 to 0.26]
Statistical Analysis 9: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.395, ANCOVA — p-value is for Interference of Pain, Relations with Others, Change; Change = Treatment + Pooled Investigator + Baseline; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.59 to 0.24]
Statistical Analysis 10: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.731, ANCOVA — p-value is for Interference of Pain, Sleep, Change; Change = Treatment + Pooled Investigator + Baseline; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.63 to 0.44]
Statistical Analysis 11: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.186, ANCOVA — p-value is for Interference of Pain, Enjoyment of Life, Change; Change = Treatment + Pooled Investigator + Baseline; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.85 to 0.17]
Statistical Analysis 12: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.220, ANCOVA — p-value is for Mean Interference Score, Change; Change = Treatment + Pooled Investigator + Baseline; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.67 to 0.16]

5. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) at Endpoint, Global Functioning Scores
Description: The SDS is completed by the patient and is used to assess the effect of the patient's symptoms on their work/social/family life. Total scores range from 0 to 30 with higher values indicating greater disruption in the patient's work/social/family life. Individual item scores range from 0-10, with higher numbers indicating greater disruption. Item 1 is for work/schoolwork, Item 2 is for social life/leisure activities, Item 3 is for family life/home responsibilities.
Time Frame: Baseline, Week 15
Population: Participants with a baseline and at least one post-baseline value.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 107 | 100
Units on a scale
  Symptoms Disrupted Work- Baseline (N=101,N=94) | 5.94 (2.01) | 5.85 (1.72)
  Symptoms Disrupted Work- Change(N=101,N=94) | -3.27 (3.06) | -2.59 (2.69)
  Symptoms Disrupted Social/Leisure - Baseline | 5.84 (1.89) | 5.73 (1.94)
  Symptoms Disrupted Social/Leisure - Change | -3.21 (2.90) | -2.60 (2.68)
  Symptoms Disrupted Family Life - Baseline | 5.50 (1.78) | 5.39 (1.83)
  Symptoms Disrupted Family Life - Change | -3.07 (2.55) | -2.45 (2.43)
  Global Functional Impairment Total Score -Baseline | 17.24 (4.58) | 17.05 (4.52)
  Global Functional Impairment Total Score -Change | -9.51 (7.56) | -7.71 (7.15)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.076, ANCOVA — p-value is for symptoms have disrupted your work/schoolwork - change; Change = Treatment + Pooled Investigator + Baseline; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-1.29 to 0.06]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.140, ANCOVA — p-value is for symptoms disrupted social/leisure - change; Change = Treatment + Pooled Investigator + Baseline; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-1.16 to 0.17]
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.087, ANCOVA — p-value is for symptoms disrupted family life - change; Change = Treatment + Pooled Investigator + Baseline; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-1.14 to 0.08]
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.083, ANCOVA — p-value is for Global Functional Impairment Total Score - change; Change = Treatment + Pooled Investigator + Baseline; Mean Difference (Final Values) = -1.62, 95% CI 2-sided [-3.46 to 0.21]

6. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) for Pain at Endpoint
Description: VAS for pain consists of 6 questions that assess overall pain, headache, back pain, shoulder pain, pain interference with daily activities, and pain while awake. Participant rates pain on a 100 millimeter (mm) line between two anchors (0= no pain and 100=very severe pain).
Time Frame: Baseline, Week 15
Population: Participants with a baseline and at least one post-baseline result within each treatment group.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 95 | 88
Units on a Scale
  Severity of Overall Pain, Past Week, Baseline | 27.56 (26.05) | 31.94 (27.62)
  Severity of Overall Pain, Past Week, Change | -15.28 (26.30) | -13.40 (29.42)
  Severity of Headaches, Past Week, Baseline | 21.11 (26.33) | 24.52 (26.68)
  Severity of Headaches, Past Week, Change | -9.44 (24.61) | -10.57 (26.36)
  Severity of Back Pain, Past Week, Baseline | 18.13 (24.99) | 17.40 (25.41)
  Severity of Back Pain, Past Week, Change | -9.40 (21.19) | -3.36 (26.55)
  Severity of Shoulder Pain, Past Week, Baseline | 16.53 (23.96) | 19.68 (27.74)
  Severity of Shoulder Pain, Past Week, Change | -8.85 (23.55) | -8.52 (27.12)
  Pain Interference, Daily Activities, Baseline | 27.19 (29.26) | 26.41 (26.03)
  Pain Interference, Daily Activities, Change | -16.92 (25.41) | -12.69 (27.53)
  Pain During Waking Hours, Past Week, Baseline | 26.84 (-28.48) | 33.22 (33.44)
  Pain During Waking Hours, Past Week, Change | -16.77 (27.53) | -14.58 (29.74)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.063, ANCOVA — p-value is for Severity of Overall Pain, Past Week, Change; Model: Change = Treatment + Pooled Investigator + Baseline; Mean Difference (Final Values) = -5.32, 95% CI 2-sided [-10.93 to 0.30]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.660, ANCOVA — p-value is for Severity of Headaches, Past Week, Change; Model: Change = Treatment + Pooled Investigator + Baseline; Mean Difference (Final Values) = -1.21, 95% CI 2-sided [-6.64 to 4.22]
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.025, ANCOVA — p-value is for Severity of Back Pain, Past Week, Change; Change = Treatment + Pooled Investigator + Baseline; Mean Difference (Final Values) = -6.03, 95% CI 2-sided [-11.30 to -0.76]
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.260, ANCOVA — p-value is for Severity of Shoulder Pain, Past Week, Change; Change = Treatment + Pooled Investigator + Baseline; Mean Difference (Final Values) = -2.93, 95% CI 2-sided [-8.06 to 2.19]
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.145, ANCOVA — p-value is for Pain Interference, Daily Activities, Change; Change = Treatment + Pooled Investigator + Baseline; Mean Difference (Final Values) = -3.67, 95% CI 2-sided [-8.61 to 1.28]
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.011, ANCOVA — p-value is for Pain During Waking Hours, Past Week, Change; Change = Treatment + Pooled Investigator + Baseline; Mean Difference (Final Values) = -7.15, 95% CI 2-sided [-12.64 to -1.66]

7. Secondary Outcome: Change From Baseline in the Hospital Anxiety and Depression Scale (HADS) Depression Subscale Score at Endpoint
Description: as for outcome 1
Time Frame: Baseline, Week 15
Population: Participants with a baseline and at least one post-baseline result within each treatment group.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 107 | 100
Units on a Scale
  Baseline | 6.90 (3.49) | 6.62 (3.35)
  Change from Baseline | -2.95 (3.82) | -1.96 (3.60)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.068, ANCOVA — p-value is for Change from Baseline; Change = Treatment + Pooled Investigator + Baseline; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-1.72 to 0.06]

ADVERSE EVENTS:
Arm/Group | Duloxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/108 | 1/102
Other Adverse Events (participants affected / at risk) | 67/108 | 45/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=108) | Placebo (N=102)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=108) | Placebo (N=102)
Palpitations (Cardiac disorders) | 3 (3) | 2 (2)
Vision blurred (Eye disorders) | 3 (3) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 7 (7) | 1 (1)
Constipation (Gastrointestinal disorders) | 10 (11) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 10 (11) | 4 (4)
Nausea (Gastrointestinal disorders) | 30 (32) | 9 (9)
Vomiting (Gastrointestinal disorders) | 6 (6) | 1 (1)
Asthenia (General disorders) | 5 (6) | 1 (1)
Fatigue (General disorders) | 4 (4) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 6 (6) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 15 (16) | 4 (4)
Headache (Nervous system disorders) | 3 (3) | 4 (4)
Somnolence (Nervous system disorders) | 12 (14) | 1 (2)
Tremor (Nervous system disorders) | 4 (4) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 5 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days